CLINICAL TRIAL: NCT01256801
Title: Gene Expression Profiling of Breast Cancer Cells in Pleural Effusion Prodict the Response of Malignant Pleural Effusion to Immunotherapy
Brief Title: Gene Expression Profiling of Breast Cancer Cells Predict the Response of Malignant Pleural Effusion
Acronym: GMPE
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Ren, Director, Peking University Cancer Hospital & Institute
Other Study IDs: GMPE
Record Dates: First submitted 2010-12-01; First posted 2010-12-09 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis; Gene Expression Profiling; Immunotherapy
Keywords: Metastatic Breast Neoplasms; Gene Expression Profiling; immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Cytokines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The cancer cells are taken from the malignant pleural effusion of breast cancer patiets.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cytokine: The patients are randomized to receive the cytokine infusion in the pleural cavity
  Interventions: Biological: cytokine

INTERVENTIONS:
Biological: cytokine — interleukin 2 2 million unit every week
  Other Names: interleukin 2 2 million unit every week

SUMMARY:
The investigators want to develop a gene expression profile for the prediction of immunotherapy response of patients with metastatic breast cancer presenting malignant pleural effusion.

DETAILED DESCRIPTION:
1. The patiets with malignant pleural effusion are randomizned to be treated with cytokins(inteleukin 2) or dendritic cells(DC) plus cytokine induced killer cells(CIK) locally.
2. Malignant pleural effusion from metastatic breast cancer patient is obtained through thoracentesis and is centrifugalized to enrich cancer cells before the therapy.
3. The enriched cancer cells are flash frozen and stored at -80℃ until processing.
4. The gene expression in pleural effusion is detected by microarray to screen gene markers that are differently expressed between groups .
5. Statistical analysis is performed using unsupervised hierarchical cluster.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be histologically confirmed with metastatic breast cancer and malignant pleural effusion
* an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* At least one measurable lesion;
* Normal cardiac, hepatic, renal and bone marrow functions;
* Life expectancy ≥3 months;
* Discontinuity of previous chemotherapy for a minimum of 4 weeks.
* Not receive chemotherapy in pleural cavity

Exclusion Criteria:

* previous history of other malignancies;
* previous surgery history on the needle biopsy organ;
* Serious or uncontrolled concurrent medical illness.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The breast cancer patiets present with pleural effusion and can receive chemotherapy.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
immunotherapy response | 1 month
  Response of malignant pleural effusion to immunotherapy is evaluated with WHO guidelines

SECONDARY OUTCOMES:
immunological status | 1 month
  compare the immunological status of pleural effusion before and after the therapy

CONTACTS AND LOCATIONS:
Overall Officials: JUN REN, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China